CLINICAL TRIAL: NCT02161666
Title: Effect of Gastric Bypass Surgery on Pancreatic Islet and Incretin Function - Follow-up Study
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Carsten Dirksen, MD, PhD, Hvidovre University Hospital
Other Study IDs: AB-CD-10-2Y
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Obesity; Gastric Bypass; Bariatric Surgery; Incretin Function; Islet Function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum specimens are retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Morbidly obese patients with normal glucose tolerance undergoing gastric bypass surgery
- Controls: Age, sex and BMI-matched healthy controls

SUMMARY:
To examine pancreatic islet function and incretin function during intravenous and oral stimulation >2 years after gastric bypass surgery in patients with normal glucose tolerance. We hypothesize that islet cell and incretin function is enhanced in response to oral, but not intravenous, stimulation - i.e. incretin released from the gut in response to oral stimulation play a key role for the enhanced islet function after gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participation in previous study (NCT01559779)

Exclusion Criteria:

* Pregnancy/lactation
* Major chronic disease develop since previous examination with possible impact on outcomes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the population undergoing gastric bypass surgery at Hvidovre Hospital (Denmark)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in islet cell function from baseline (preoperatively) | >24 months
  Change in insulin and glucagon secretion during oral and intravenous stimulation after gastric bypass

SECONDARY OUTCOMES:
Change in glucose tolerance during oral glucose tolerance test | >24 months
  Fasting, peak and nadir glucose during oral glucose tolerance test
Arterio-venous glucose difference during oral glucose tolerance test after gastric bypass | >24 months
  Differences in arterial and venous plasma glucose during oral glucose stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, MD, PhD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Danmark, Denmark

REFERENCES:
- [Derived] Dirksen C, Eiken A, Bojsen-Moller KN, Svane MS, Martinussen C, Jorgensen NB, Holst JJ, Madsbad S. No Islet Cell Hyperfunction, but Altered Gut-Islet Regulation and Postprandial Hypoglycemia in Glucose-Tolerant Patients 3 Years After Gastric Bypass Surgery. Obes Surg. 2016 Sep;26(9):2263-2267. doi: 10.1007/s11695-016-2197-x. PMID 27138601